CLINICAL TRIAL: NCT01145131
Title: Dietary Interventions for Muscle Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MEC 10-3-065
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Aging
Keywords: muscle; FSR; protein; meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beef steak (Experimental)
  Interventions: Other: Intact or minced beef meat
- Minced beef (Experimental)
  Interventions: Other: Intact or minced beef meat

INTERVENTIONS:
Other: Intact or minced beef meat — 135 gram piece of intact or minced beef meat, beef steak or minced beef resp.
  Other Names: Beef steak; Minced beef; Beef patty; Steak; Hamburger; Ground beef

SUMMARY:
Dietary intervention to prevent sarcopenia in elderly people. The objective of this study is to test whether meat structure plays an important role in protein digestion, to maximise the amino acid availability and to stimulate the muscle protein growth in elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese male subjects (BMI<30) between the age of 65-85 years.

Exclusion Criteria:

* Type II diabetes or other known diseases, use of medication, female, other ages or BMI than indicated above, participation in any regular exercise program.

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | 6 h postprandial period
  Muscle protein synthesis will be expressed as fractional synthetic rate (FSR) by dividing the increment in enrichment in the product, i.e. protein-bound D5phe tracer, by the enrichment of the precursor (=plasma availability).

SECONDARY OUTCOMES:
Dietary amino acid plasma availability | 6h postprandial period
  The exogenous rate of phenylalanine appearance will be used to assess the bio-availability of dietary-protein derived amino acids in the circulation during the 6h postprandial period following meat intake

CONTACTS AND LOCATIONS:
Overall Officials: B Pennings, Ir, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Universiteit Maastricht, Bewegingswetenschappen, Maastricht, Limburg, Netherlands

REFERENCES:
- [Result] Mioche L, Bourdiol P, Monier S, Martin JF, Cormier D. Changes in jaw muscles activity with age: effects on food bolus properties. Physiol Behav. 2004 Sep 30;82(4):621-7. doi: 10.1016/j.physbeh.2004.05.012. PMID 15327909
- [Result] Mioche L, Bourdiol P, Monier S. Chewing behaviour and bolus formation during mastication of meat with different textures. Arch Oral Biol. 2003 Mar;48(3):193-200. doi: 10.1016/s0003-9969(03)00002-5. PMID 12648556
- [Derived] Pennings B, Groen BB, van Dijk JW, de Lange A, Kiskini A, Kuklinski M, Senden JM, van Loon LJ. Minced beef is more rapidly digested and absorbed than beef steak, resulting in greater postprandial protein retention in older men. Am J Clin Nutr. 2013 Jul;98(1):121-8. doi: 10.3945/ajcn.112.051201. Epub 2013 May 1. PMID 23636241
- See also: Information about research performed by the Maastricht Muscle Metabolism group at MUMC — http://www.m3-research.nl